CLINICAL TRIAL: NCT04945486
Title: The Effect of a Peer-mentor Intervention on Inequality in Cardiac Rehabilitation Attendance: a Mixed Method Intervention Study Among Older Vulnerable Patients With Ischemic Heart Disease
Brief Title: The Effect of Peer-mentor Support for Older Vulnerable Patients With Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Copenhagen (Other)
Collaborators: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Maria Kjøller Pedersen, Associate Professor, University College Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Alias: 200348 RCT
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Masking Description: Masking is not possible
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-mentoring (Experimental): The patients (mentees) are matched with a peer-mentor i.e. a person with a similar life situation or health problem as one self
  Interventions: Other: Peer-mentor intervention
- Usual care (No Intervention): Usual care provided by professional healthcare workers

INTERVENTIONS:
Other: Peer-mentor intervention — Peer-mentor support for up to 6 months
  Arms: Peer-mentoring

SUMMARY:
BACKGROUND: Advanced treatment regimens have reduced cardiovascular mortality resulting in an increasingly older Ischemic Heart Disease (IHD) population in need of cardiac rehabilitation (CR) , the majority (74%) is above 60 years. The positive effect of CR is well established; CR reduces cardiovascular mortality, lowers hospital admissions, and improves quality of life among patients with IHD. These positive effects of CR has also been established among older patients. The inherent problem lies in the low attendance rate, often below 50%. Several studies, including studies from Denmark, have shown that low participation in CR is most prevalent among older, vulnerable and female patients. The notion vulnerable covers patients with low socioeconomic position (SEP), patients with non-western background and patients living alone, as these groups have particularly low CR attendance. Effective interventions aiming at increasing CR attendance among these low attending groups are thus warranted and the current study will seek to address this.

AIM: To test the effect of a peer-mentor intervention among older vulnerable IHD patients.

DESIGN AND METHODS: The study is designed as a two arm RCT-study applying mixed methods.

Power calculations were based upon primary outcome 'Cardiac rehabilitation (CR) attendance'. Proportion attending CR in control group was set at 25% and intervention group at 50% based upon previous research. With a 5% significance level and 80% power. 110 patients were required (55 in each group) to have a 80% chance of detecting, as significant at the 5% level, an increase in the primary outcome measure from 25% in the control group to 50% in the experimental group.

Expected dropout was 6%. I.e., in total 117 patients are enrolled.

Patients (n=117) are recruited by a dedicated research nurse before discharge from the cardiology department at Nordsjællands Hospital and randomized (with 1:1 individual randomisation) to peer-mentor intervention or usual care. Data is collected through both qualitative and quantitative data (mixed methods). Data is collected at three timepoints, baseline, 12 weeks and 24 weeks. The patients (mentees) are matched with peer-mentors. Peer-mentoring (i.e. mentoring by a person with a similar life situation or health problem as one self) is a low-cost intervention that holds the potential to improve CR attendance and improve physical and psychological outcomes among older patients. Peer-mentors are role models who can guide and support patients overcoming barriers of CR attendance. Peer-mentoring is unexplored in a CR setting among older, female and vulnerable IHD patients; establishing the novelty of the current study.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years and diagnosed with IHD and referred to CR and female or low SEP or single living or non-western background

Exclusion Criteria:

* Patients unable to provide written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Cardiac rehabilitation attendance | 24 weeks
  Measured as 'self-reported CR attendance'

SECONDARY OUTCOMES:
Change in Health-related Quality of Life | Baseline to 24 weeks
  Measured using the 'HeartQoL' 'Health-related Quality of Life Questionnaire'. Min. score: 0, max score: 42. Higher scores indicating a better outcome.
Change in Self-efficacy | Baseline to 24 weeks
  Measured using the questionnaire 'General self-efficacy scale'. Min score: 10, max score: 40. Higher scores indicating a better outcome
Change in symptoms of anxiety and depression | Baseline to 24 weeks
  Measured using the questionnaire 'The hospital anxiety and depression scale' (HADS). Min. score: 0, max score 42. Lower scores indicating a better outcome
Change in dietary quality | Baseline to 24 weeks
  Measured using the questionnaire 'Heartdiet'. Higher scores indicating a better outcome
Change in physical activity | Baseline to 24 weeks
  Measured using the questionnaire 'Heartdiet'. Higher scores indicating a better outcome
Qualitative content of disease trajectory | Baseline to 24 weeks
  Semi-structured qualitative interviews with patients (n=20-25)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital - Frederikssund, Frederikssund
  - Nordsjællands Hospital - Hillerød, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen M, Petersen RA, Boateng T, Egerod I, Overgaard D, Bennich BB. Peer-Mentor Support for Older, Vulnerable Patients With Ischemic Heart Disease: A Mixed Methods Process-Outcome Evaluation. J Adv Nurs. 2025 Dec;81(12):8946-8958. doi: 10.1111/jan.16899. Epub 2025 Mar 17. PMID 40095257